CLINICAL TRIAL: NCT00818233
Title: Intra-observer and Inter-observer Variability With Dynamic Contour Tonometry.
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty recruiting patients. PI left research facility.
Sponsor: Yale University (Other)
Responsible Party: Hylton R. Mayer, Yale University
Other Study IDs: 0601001047
Record Dates: First submitted 2008-11-18; First posted 2009-01-07 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Intraocular Pressure
Keywords: dynamic contour tonometry; variability; pulse amplitude; Ocular pulse amplitude

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observation: Variability will be assessed between each examiner.
  Interventions: Device: Dynamic contour tonometry

INTERVENTIONS:
Device: Dynamic contour tonometry — Observe variability of measurements by dynamic contour tonometry
  Other Names: PASCAL tonometry; DCT

SUMMARY:
The aim of the protocol is to document intra-observer and inter-observer variability with dynamic contour tonometry, and will also test the theory that pulse amplitude, as measured by dynamic contour tonometry, is correlated with the difference in systolic and diastolic blood pressures.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy eyes
* Minimal to moderate refractive error
* Willingness to participate in the study

Exclusion Criteria:

* Diagnosis of any type of glaucoma
* Any prior ocular surgery
* Any prior ocular trauma
* Any known anterior segment pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, competent adults with normal, healthy eyes.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-01

PRIMARY OUTCOMES:
The variability of intraocular pressure measurements using dynamic contour tonometry | Same day

SECONDARY OUTCOMES:
Observe how pulse amplitude, as measured by dynamic contour tonometry, correlates with the difference in systolic and diastolic blood pressures | Same day

CONTACTS AND LOCATIONS:
Overall Officials: Hylton R Mayer, MD, Principal Investigator — Yale University
Locations (1):
- Yale Eye Center, New Haven, Connecticut, United States